CLINICAL TRIAL: NCT00827931
Title: Prospective Randomized Phase IV Open Label Comparative Study Of Tranexamic Acid Plus Standard Of Care Vs Standard Of Care For The Reduction Of Blood Loss In Patients Undergoing Major Abdominal Surgery
Brief Title: Study Of Tranexamic Acid For The Reduction Of Blood Loss In Patients Undergoing Major Abdominal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B1461001
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Results first posted 2012-04-26 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Biliary Tract Surgical Procedures; Pancreaticoduodenectomy; Esophagectomy; Colectomy; Gastrectomy
Keywords: tranexamic acid; major abdominal surgery; blood loss
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): end of the operation and on the mornings of the first, second, fourth and seventh postoperative days.
  Interventions: Drug: Tranexamic acid + Standard of Care
- B (Other): Standard of Care
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Drug: Tranexamic acid + Standard of Care — Tranexamic acid given slowly intravenously (15 mg/kg body weight) 15 minutes before surgery followed by a second dose at three hour interval from first dose and third dose at three hour interval from the second + standard of care (Standard of care includes the routine surgical and anesthetic techniques being utilized to control blood loss)
  Arms: A
Procedure: Standard of Care — Standard of care includes the routine surgical and anesthetic techniques being utilized to control blood loss
  Arms: B

SUMMARY:
Tranexamic acid has been shown to reduce postoperative blood losses and transfusion requirements in various types of major surgery (orthopedic surgery, spine surgery, cardiopulmonary bypass, liver resections, and gynecological cancers).The current trial is being conducted to compare the efficacy of tranexamic acid plus standard of care versus standard of care in reduction of blood loss in patients undergoing major abdominal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing major abdominal surgery (Biliary strictures, Pancreatico-duodenectomy, Esophagectomy, Total proctocolectomy, Hemicolectomy, Gastrectomy, Other major abdominal surgeries with similar expected blood loss)

Exclusion Criteria:

* Patients with a platelet count less than 100, 000/mm3 or history of thrombocytopenia.
* Patients with known coagulopathy.
* Patients with anemia (hemoglobin levels less than 8 mg/dl)
* Patients with documented DVT or PE at screening or in past three months.
* Patients with any associated major illness (e.g., severe cardiac or respiratory disease).
* Anticoagulants (other than LMWH or heparin in prophylactic doses to prevent deep vein thrombosis), direct thrombin inhibitors or thrombolytic therapy administered or completed within last week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- India (2):
  - Pfizer Investigational Site, Surat, Gujarat
  - Pfizer Investigational Site, Vadodara, Gujarat

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1461001&StudyName=Study%20Of%20Tranexamic%20Acid%20For%20The%20Reduction%20Of%20Blood%20Loss%20In%20Patients%20Undergoing%20Major%20Abdominal%20Surgery

RESULTS

PARTICIPANT FLOW:
Groups:
- Tranexamic Acid Plus Standard of Care: Tranexamic acid given slowly intravenously (IV) (15 milligram (mg)/kilogram (kg) body weight) 15 minutes before surgery followed by a second dose at 3 hour interval from first dose and third dose at 3 hour interval from the second + Standard of care (included the routine surgical and anesthetic techniques being utilized to control blood loss).
- Standard of Care: Standard of care included the routine surgical and anesthetic techniques being utilized to control blood loss.
Period: Overall Study
Arm/Group | Tranexamic Acid Plus Standard of Care | Standard of Care
Started | 49 | 45
Completed | 43 | 39
Not Completed | 6 | 6
Not completed — Death | 3 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid Plus Standard of Care | Standard of Care | Total
Number analyzed (Participants) | 49 | 45 | 94
Age, Customized [Number; unit: Participants]
  18 to 44 years | 24 | 16 | 40
  45 to 64 years | 21 | 22 | 43
  Greater than or equal to 65 years | 4 | 7 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 33 | 29 | 62

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Blood Loss
Description: Post-operative blood loss was defined as the sum of the drainage volumes measured over post-operative days 1, 2, and at drain removal. It was measured by weighing the drapes/ dressings or swabs prior to soaking to measure difference in weight and checking drain collectors until drains were removed.
Time Frame: Post-operation, Day 1, Day 2 up to drain removal
Population: Full Analysis Set (FAS) population included all randomized participants in compliance with the intent-to-treat analysis principle. Participants who had no post-baseline data for a given endpoint was not included in the analysis of that endpoint.
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | Tranexamic Acid Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 23 | 21
milliliter (mL) | 394.3 (366.36) | 494.3 (503.94)
Statistical Analysis 1: Comparison: Tranexamic Acid Plus Standard of Care vs Standard of Care; The null hypothesis applicable to the efficacy analyses was that there was no difference between tranexamic acid plus standard care compared to standard care alone. The alternative hypothesis was that there was a difference; Test type: Superiority or Other; p = 0.460, t-test, 2 sided; Mean Difference (Final Values) = -99.9, 95% CI 2-sided [-371.4 to 171.5], Standard Error of Mean 131.99

2. Secondary Outcome: Intra-operative Blood Loss
Description: Intra-operative blood loss was measured by weighing the drapes/ dressings or swabs prior to soaking to measure difference in weight and checking drain collectors until drains were removed.
Time Frame: Day 1 (End of surgery)
Population: FAS population included all randomized participants in compliance with the intent-to-treat analysis principle. Participants who had no post-baseline data for a given endpoint was not included in the analysis of that endpoint.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tranexamic Acid Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 23 | 21
mL | 599.2 (419.58) | 682.8 (555.52)
Statistical Analysis 1: Comparison: Tranexamic Acid Plus Standard of Care vs Standard of Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.579, t-test, 2 sided; Mean Difference (Final Values) = -83.6, 95% CI 2-sided [-386.5 to 219.3], Standard Error of Mean 147.61

3. Secondary Outcome: Total Blood Loss
Description: Total blood loss was defined as the sum of intra-operative and post-operative blood loss. It was measured by weighing the drapes/ dressings or swabs prior to soaking to measure difference in weight and checking drain collectors until drains were removed.
Time Frame: Baseline through Day 2 post-surgery
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tranexamic Acid Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 23 | 21
mL | 993.6 (703.63) | 1177.1 (879.94)
Statistical Analysis 1: Comparison: Tranexamic Acid Plus Standard of Care vs Standard of Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.452, t-test, 2 sided; Mean Difference (Final Values) = -183.5, 95% CI 2-sided [-672.6 to 305.5], Standard Error of Mean 239.19

4. Secondary Outcome: Total Blood Loss as Assessed by the Gross' Formula
Description: Gross' formula for estimating total blood loss: Estimated blood volume multiplied by (*) [(hematocrit initial minus hematocrit final) divided by hematocrit average]; where estimated blood volume equals body weight in kilograms (kg) *70 mL/kg.
Time Frame: Baseline through Day 2 post-surgery
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tranexamic Acid Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 23 | 21
mL | 17.8 (451.24) | 435.5 (558.74)
Statistical Analysis 1: Comparison: Tranexamic Acid Plus Standard of Care vs Standard of Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.010, t-test, 2 sided; Mean Difference (Final Values) = -417.7, 95% CI 2-sided [-729.4 to -106.1], Standard Error of Mean 152.51

5. Secondary Outcome: Percentage of Participants Receiving Transfusions
Description: A uniform transfusion protocol was maintained for all participants in the study. Transfusion to be triggered at 8.0 milligram/deciliter (mg/dL) hemoglobin or hematocrit value of 24 percent.
Time Frame: Up to Day 7 post-surgery
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tranexamic Acid Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 23 | 21
Percentage of participants | 21.7 [7.5 to 43.7] | 14.3 [3.0 to 36.3]
Statistical Analysis 1: Comparison: Tranexamic Acid Plus Standard of Care vs Standard of Care; Fisher's exact test was used at 5% level of significance; Test type: Superiority or Other; p = 0.701, Fisher Exact

6. Secondary Outcome: Hemoglobin Levels
Time Frame: End of surgery, Day 1, Day 2, Day 4 and Day 7/End of treatment (EoT) post-surgery
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Gram/Deciliter (g/dL)
Arm/Group | Tranexamic Acid Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 23 | 21
Gram/Deciliter (g/dL)
  End of surgery | 11.6 (2.16) | 12.1 (1.30)
  Day 1 | 11.3 (1.44) | 11.6 (1.41)
  Day 2 | 10.4 (1.70) | 11.0 (1.41)
  Day 4 | 10.8 (1.67) | 10.9 (1.39)
  Day 7/EoT | 11.0 (1.38) | 11.1 (1.60)

7. Secondary Outcome: Number of Participants With Deep Vein Thrombosis (DVT) Post Surgery
Description: DVT was defined if a segment of the deep vein of the lower limb was not compressible or a previous compressive vein became non compressive or there was no flow in the underlying vessel. Symptoms of DVT included pain in the lower limb, localized tenderness, swelling and warmth.
Time Frame: Day 7 post-surgery
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Tranexamic Acid Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 23 | 21
Participants | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Tranexamic Acid Plus Standard of Care | Standard of Care
Serious Adverse Events (participants affected / at risk) | 9/49 | 7/45
Other Adverse Events (participants affected / at risk) | 22/49 | 14/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tranexamic Acid Plus Standard of Care (N=49) | Standard of Care (N=45)
Bradycardia (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 2 | 3
Myocardial infarction (Cardiac disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Biliary tract disorder (Hepatobiliary disorders) | 1 | 1
Infectious peritonitis (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Suture rupture (Injury, poisoning and procedural complications) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tranexamic Acid Plus Standard of Care (N=49) | Standard of Care (N=45)
Anaemia (Blood and lymphatic system disorders) | 5 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 1
Abscess (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 0
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 4 | 4
Blood glucose increased (Investigations) | 0 | 1
Blood pressure decreased (Investigations) | 1 | 2
Haematocrit decreased (Investigations) | 1 | 3
Haemoglobin decreased (Investigations) | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Bradykinesia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria contact (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 4 | 1

LIMITATIONS AND CAVEATS:
The intended FAS population was planned to include participants from 2 sites, however due to non-reliability of data from one of the sites, the actual FAS population included participants from a single site only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.